CLINICAL TRIAL: NCT06321237
Title: Effect of Ear Vagus Nerve Stimulator on Symptom Improvement and Intestinal Microbiome in Patients With Irritable Bowel
Brief Title: Influence of Ear Vagus Nerve Stimulator on Patients With IBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huaping Xie (Other)
Responsible Party: Sponsor-Investigator, Huaping Xie, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TJ-IRB202402130
Record Dates: First submitted 2024-03-11; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Ear nail stimulator; Gut microbiota; Vagus nerve stimulation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The true-true stimulus group (Active Comparator): During the 8-week intervention, the patient used the ear nail stimulator to give true stimulation, that is, the vagus nerve stimulation with a pulse width of 200μs and a frequency of 30Hz
  Interventions: Device: Vagus nerve stimulation for 8 weeks
- The true-false stimulus group (Experimental): During the 8-week intervention, the first 4 weeks of the auricular stimulator used by the patient were given true stimulation, that is, vagus nerve stimulation with a pulse width of 200μs and a frequency of 30Hz; The next 4 weeks were given as false stimuli
  Interventions: Device: Vagus nerve stimulation for the first 4 weeks
- The false-true stimulus group (Experimental): During the 8-week intervention, the first 4 weeks of the patient's ear nail stimulator gave false stimulation; The stimulation given in the last 4 weeks is true stimulation, that is, vagus nerve stimulation with pulse width of 200μs and frequency of 30Hz
  Interventions: Device: Vagus nerve stimulation for the last 4 weeks
- The false-false stimulus group (Placebo Comparator): Over the course of the 8-week intervention, the patient used an ear nail stimulator that gave false stimulation
  Interventions: Device: Pseudostimulus

INTERVENTIONS:
Device: Vagus nerve stimulation for 8 weeks — The vagus nerve at the position of the ear nail was stimulated by an ear nail stimulator with pulse width of 200μs and frequency of 30Hz in patients with IBS for 8 weeks
  Arms: The true-true stimulus group
Device: Vagus nerve stimulation for the first 4 weeks — The vagus nerve at the position of the ear nail was stimulated by an ear nail stimulator with pulse width of 200μs and frequency of 30Hz in patients with IBS for the first 4 weeks
  Arms: The true-false stimulus group
Device: Vagus nerve stimulation for the last 4 weeks — The vagus nerve at the position of the ear nail was stimulated by an ear nail stimulator with pulse width of 200μs and frequency of 30Hz in patients with IBS for the last 4 weeks
  Arms: The false-true stimulus group
Device: Pseudostimulus — The patient is given some electrical stimulation but not vagus nerve stimulation
  Arms: The false-false stimulus group

SUMMARY:
Irritable bowel syndrome (IBS) is a very common functional digestive disorder characterized by chronic abdominal pain and altered bowel habits in the absence of biological or structural abnormalities. In the field of IBS, effective drug treatments are very limited, and patients are urgently looking for alternatives, including probiotics, hypnotherapy, osteopathy, dietary changes, and fecal microbiota transplants. In recent years, with the continuous elucidation of vagus nerve mechanisms, IBS patients are increasingly interested in bioelectrical regulation, and these patients are often skeptical of traditional drug treatment and believe that drugs are prone to side effects. For several reasons, vagus nerve stimulation (VNS) may be a promising option for improving IBS symptoms. In this experiment, the portable ear nail stimulator produced by Ruishen Medical can accurately stimulate the ear nail, transdermal stimulation of the ear vagus nerve, and give full play to its therapeutic effect. Therefore, the purpose of this clinical trial is to use ear nail stimulator in patients with IBS to explore whether it has therapeutic effects on patients with IBS. To explore the influence of tVNS therapy on irritable bowel syndrome compared with drug therapy, it is hoped that the use of TVNS therapy can reduce the use of related drugs, or even replace drugs. This study intends to recruit a group of patients with irritable bowel syndrome to use the portable ear nail stimulator, (1) to observe whether the symptoms of irritable bowel syndrome patients are improved; (2) To analyze the changes of intestinal microbes in patients with IBS; (3) Verify whether the level of intestinal inflammation is reduced and discover metabolic markers in the intestine.

DETAILED DESCRIPTION:
The human gut microbiome is one of the most densely populated microbial communities on Earth and contains highly diverse microbial communities that provide metabolic, immune and protective functions and play a critical role in human health. The gastrointestinal microbiota is influenced by a variety of factors, including neurological stress, genetics, host physiology (host age, disease, etc.), and environmental factors such as living conditions and drug use. At the same time, the vagus nerve (VN) is considered a key component of the autonomic nervous system (ANS), which innervates most of the digestive tract and many gastrointestinal organs such as the esophagus, stomach, small intestine, and colon, as well as vital organs such as the liver, pancreas, and gallbladder in the digestive system. The vagus nerve transmits excitement to the corresponding brain region by sensing intestinal stimulation, and regulates the gut and brain bidirectionally through the "gut-brain axis". Recent studies have shown that VN has anti-inflammatory effects. This vagus function is mediated through a variety of pathways, some of which remain controversial. The first is the anti-inflammatory pathway of the hypothalamic-pituitary-adrenal axis, stimulated by the afferent fibers of the vagus nerve, where the adrenal glands release cortisol, which provides an important first innate defense against inflammatory infections and helps restore homeostasis in the body. The second, known as the cholinergic anti-inflammatory pathway, releases acetylcholine (ACh) at the synaptic junction with macrophages through the vagal efferent fibre-mediated synaptic connections of intestinal neurons. Acetylcholine binds to the α-7-nicotinic acetylcholine receptor of macrophages and inhibits the release of tumor necrosis (TNF)α, a pro-inflammatory cytokine. The final pathway is the splenic sympathetic anti-inflammatory pathway, where VN stimulates the splenic sympathetic nerve to release acetylcholine from norepinephrine (norepinephrine) at the distal end. Finally, ACh inhibits the release of TNF-α from splenic macrophages through the α-7-nicotinic ACh receptor. Irritable bowel syndrome (IBS) is a very common functional digestive disorder characterized by chronic abdominal pain and altered bowel habits in the absence of biological or structural abnormalities. In the field of IBS, effective drug treatments are very limited, and patients are urgently looking for alternatives, including probiotics, hypnotherapy, osteopathy, dietary changes, and fecal microbiota transplants. In recent years, with the continuous elucidation of vagus nerve mechanisms, IBS patients are increasingly interested in bioelectrical regulation, and these patients are often skeptical of traditional drug treatment and believe that drugs are prone to side effects. For several reasons, vagus nerve stimulation (VNS) may be a promising option for improving IBS symptoms. Vagus nerve stimulation (VNS) is currently used as a treatment option for many clinical conditions, such as heart failure, migraines, and inflammatory bowel disease. VNS techniques are mainly divided into invasive (surgical implantation) and non-invasive (percutaneous)VNS techniques. Invasive VNS (iVNS) involve implanting a programmable pulse generator device in the chest wall and placing electrodes around the left (typical) cervical vagus nerve. As it stands, iVNS has several potential risks, such as bradycardia and cardiac arrest, and localized infections around the wound. The transcutaneous VNS (tVNS) delivery system relies on the skin distribution of the afferent nerve of the vagus nerve to intervene in the outer ear (the auricular branch of the vagus nerve) or the neck (the cervical branch of the vagus nerve), thereby avoiding the risk of surgical implantation of the VNS delivery device and promoting further research on the application of tVNS. In this experiment, the portable ear nail stimulator produced by Ruishen Medical can accurately stimulate the ear nail, transdermal stimulation of the ear vagus nerve, and give full play to its therapeutic effect. Therefore, the purpose of this clinical trial is to use ear nail stimulator in patients with IBS to explore whether it has therapeutic effects on patients with IBS. To explore the influence of tVNS therapy on irritable bowel syndrome compared with drug therapy, it is hoped that the use of TVNS therapy can reduce the use of related drugs, or even replace drugs. This study intends to recruit a group of patients with IBS to use the portable ear nail stimulator. The purpose of the study is (1) to observe whether the symptoms of IBS patients are improved; (2) To analyze the changes of intestinal microbes in patients with IBS; (3) Verify whether the level of intestinal inflammation is reduced and discover metabolic markers in the intestine. This was a randomized, double-blind study with no placebo group and enrolled 40 patients diagnosed with diarrheal irritable bowel syndrome. The enrolled patients were randomly assigned to tVNS true stimulation (real transcutaneous vagal stimulation) and false stimulation (same instrument but no vagal stimulation) at different times. This study does not require recruitment advertisements, and subjects are recruited on a completely voluntary basis. Possible risks during the experiment are explained to subjects and informed consent is signed after they agree to join the study. The volunteers who agreed to join the experiment were surveyed by questionnaire to obtain their intestinal health and other health conditions, and screened according to the above research object selection criteria and exclusion criteria. The collected samples are named by number, which will not disclose the personal information of the subjects. The identity of the subjects is kept secret throughout the study process, and only the number and disease phenotype are visible. Subjects may withdraw from the study at any time. This study will analyze the composition and structure of the gut microbiota of the subjects, and the subjects can keep abreast of the progress of the testing and analysis and obtain their own relevant data. In this study, the Ruishenan auricular vagus nerve stimulator is used directly without installation. Easy to carry, can be opened at any time stimulation, does not affect daily work and life. Currently approved indications are: adjuvant therapy for sleep disorders, anxiety, loss of appetite, fatigue, and adjuvant therapy for diabetes. In this study, ear nail stimulation with a pulse width of 200μs and a frequency of 30Hz was used for 3 hours a day for 8 weeks to improve the clinical symptoms of patients with irritable bowel syndrome. The experimental plan was to collect stool samples from the recruited patients with diarrheal irritable bowel syndrome, and use the ear conchal stimulator for 3h every day with pulse width of 200μs and frequency of 30Hz. The treatment lasted for 8 weeks [28], and each patient was randomly selected as true or false stimulus every 4 weeks, and a total of 4 groups were generated, namely true-true, true-false, false-true, and false-false (Figure 2). The volunteers' stool samples were collected on days 0, 28 and 56. Stool samples were collected two weeks after treatment. On day 0 and every 7 days thereafter, the patients filled in the questionnaire, and a total of 11 questionnaires were collected.

ELIGIBILITY:
Inclusion Criteria:

1、All patients were excluded from colorectal tumors by colonoscopy within two years, and their clinical manifestations were diarrheal irritable bowel syndrome, which met the diagnostic criteria of Rome IV

Exclusion Criteria:

1. Colonoscopy excludes patients with colorectal tumors within one or two years
2. Patients with other gastrointestinal disorders
3. Patients with a history of prior abdominal surgery, cardiovascular disease, or serious illness
4. In the past month, participants had used drugs that could have affected the study results (e.g., probiotics, prebiotics, antibiotics, laxatives, motility agents).
5. Patients participating in other clinical studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-26 (Estimated); Study Completion 2024-06-09 (Estimated)

PRIMARY OUTCOMES:
Changes in irritable bowel symptoms | 90 days
  Changes in irritable bowel were evaluated by pain degree, frequency of diarrhea, and degree of abdominal distension. Pain degree refers to the use of psychometric practice to evaluate patients' subjective feelings, which is also considered to be a major factor in the evaluation of health-related poor quality of life (HRQL). We measured the severity of IBS using the Gastrointestinal Symptom Score Scale (GSRS-IBS) for IBS. On the GSRS-IBS scale, a score of 1 to 3 is defined as mild, a score of 4 or 5 is defined as more severe, and a score of 6 or 7 is defined as particularly severe
Changes in the diversity of intestinal flora | 90 days
  The changes of intestinal flora diversity before and after the use of ear nail stimulator were analyzed.Alpha diversity is a combination of species richness and evenness in a designated ecosystem. the Bray-Curtis distance reflects the variability in community composition and structure, with greater distances resulting in greater variability between communities.
Changes in the relative abundance of species of intestinal flora | 90 days
  To analyse the changes of relative abundance of species before and after the use of ear nail stimulator in patients.According to the species abundance table of each species, Krona analysis, relative abundance profile display,relative abundance cluster thermogram display, PCA and PCoA dimension reduction analysis, and Wilcoxon test of different species between groups were carried out.
Changes in the number of intestinal flora | 90 days
  Analyse the changes in the number of fecal flora before and after the use of ear nail stimulator in patients with constipation. In order to demonstrate more visually the changes in flora abundance after administration of resistant starch, statistical analyses were carried out using the number of patients who had a 1.5-fold increase or decrease in intestinal flora abundance before and after administration of resistant starch in all patients

CONTACTS AND LOCATIONS:
Overall Officials: ping h Xie, Study Chair — Tongji Medical College of Huazhong University of Science and Technology; qiang Ding, Principal Investigator — Tongji Medical College of Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No
Questionnaires filled out by patients before and after using ear nail stimulator, and metagenomic sequencing results of stool samples

REFERENCES:
- [Result] Jumpertz R, Le DS, Turnbaugh PJ, Trinidad C, Bogardus C, Gordon JI, Krakoff J. Energy-balance studies reveal associations between gut microbes, caloric load, and nutrient absorption in humans. Am J Clin Nutr. 2011 Jul;94(1):58-65. doi: 10.3945/ajcn.110.010132. Epub 2011 May 4. PMID 21543530
- [Result] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Result] Goldsmith JR, Sartor RB. The role of diet on intestinal microbiota metabolism: downstream impacts on host immune function and health, and therapeutic implications. J Gastroenterol. 2014 May;49(5):785-98. doi: 10.1007/s00535-014-0953-z. Epub 2014 Mar 21. PMID 24652102
- [Result] Bonaz B, Sinniger V, Pellissier S. Anti-inflammatory properties of the vagus nerve: potential therapeutic implications of vagus nerve stimulation. J Physiol. 2016 Oct 15;594(20):5781-5790. doi: 10.1113/JP271539. Epub 2016 May 1. PMID 27059884
- [Result] Yu CD, Xu QJ, Chang RB. Vagal sensory neurons and gut-brain signaling. Curr Opin Neurobiol. 2020 Jun;62:133-140. doi: 10.1016/j.conb.2020.03.006. Epub 2020 May 4. PMID 32380360
- [Result] Johnston GR, Webster NR. Cytokines and the immunomodulatory function of the vagus nerve. Br J Anaesth. 2009 Apr;102(4):453-62. doi: 10.1093/bja/aep037. Epub 2009 Mar 3. PMID 19258380
- [Result] Pavlov VA, Wang H, Czura CJ, Friedman SG, Tracey KJ. The cholinergic anti-inflammatory pathway: a missing link in neuroimmunomodulation. Mol Med. 2003 May-Aug;9(5-8):125-34. PMID 14571320
- [Result] Matteoli G, Gomez-Pinilla PJ, Nemethova A, Di Giovangiulio M, Cailotto C, van Bree SH, Michel K, Tracey KJ, Schemann M, Boesmans W, Vanden Berghe P, Boeckxstaens GE. A distinct vagal anti-inflammatory pathway modulates intestinal muscularis resident macrophages independent of the spleen. Gut. 2014 Jun;63(6):938-48. doi: 10.1136/gutjnl-2013-304676. Epub 2013 Aug 8. PMID 23929694
- [Result] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Result] Wang Y, Zheng F, Liu S, Luo H. Research Progress in Fecal Microbiota Transplantation as Treatment for Irritable Bowel Syndrome. Gastroenterol Res Pract. 2019 Dec 1;2019:9759138. doi: 10.1155/2019/9759138. eCollection 2019. PMID 31885549
- [Result] Shah K, Ramos-Garcia M, Bhavsar J, Lehrer P. Mind-body treatments of irritable bowel syndrome symptoms: An updated meta-analysis. Behav Res Ther. 2020 May;128:103462. doi: 10.1016/j.brat.2019.103462. Epub 2019 Nov 12. PMID 32229334
- [Result] Muller A, Franke H, Resch KL, Fryer G. Effectiveness of osteopathic manipulative therapy for managing symptoms of irritable bowel syndrome: a systematic review. J Am Osteopath Assoc. 2014 Jun;114(6):470-9. doi: 10.7556/jaoa.2014.098. PMID 24917634
- [Result] Ford AC, Harris LA, Lacy BE, Quigley EMM, Moayyedi P. Systematic review with meta-analysis: the efficacy of prebiotics, probiotics, synbiotics and antibiotics in irritable bowel syndrome. Aliment Pharmacol Ther. 2018 Nov;48(10):1044-1060. doi: 10.1111/apt.15001. Epub 2018 Oct 8. PMID 30294792
- [Result] Bonaz B, Picq C, Sinniger V, Mayol JF, Clarencon D. Vagus nerve stimulation: from epilepsy to the cholinergic anti-inflammatory pathway. Neurogastroenterol Motil. 2013 Mar;25(3):208-21. doi: 10.1111/nmo.12076. Epub 2013 Jan 29. PMID 23360102
- [Result] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Result] Bonaz B, Bazin T, Pellissier S. The Vagus Nerve at the Interface of the Microbiota-Gut-Brain Axis. Front Neurosci. 2018 Feb 7;12:49. doi: 10.3389/fnins.2018.00049. eCollection 2018. PMID 29467611
- [Result] Foster JA, Rinaman L, Cryan JF. Stress & the gut-brain axis: Regulation by the microbiome. Neurobiol Stress. 2017 Mar 19;7:124-136. doi: 10.1016/j.ynstr.2017.03.001. eCollection 2017 Dec. PMID 29276734
- [Result] De Ferrari GM, Crijns HJ, Borggrefe M, Milasinovic G, Smid J, Zabel M, Gavazzi A, Sanzo A, Dennert R, Kuschyk J, Raspopovic S, Klein H, Swedberg K, Schwartz PJ; CardioFit Multicenter Trial Investigators. Chronic vagus nerve stimulation: a new and promising therapeutic approach for chronic heart failure. Eur Heart J. 2011 Apr;32(7):847-55. doi: 10.1093/eurheartj/ehq391. Epub 2010 Oct 28. PMID 21030409
- [Result] Botha C, Farmer AD, Nilsson M, Brock C, Gavrila AD, Drewes AM, Knowles CH, Aziz Q. Preliminary report: modulation of parasympathetic nervous system tone influences oesophageal pain hypersensitivity. Gut. 2015 Apr;64(4):611-7. doi: 10.1136/gutjnl-2013-306698. Epub 2014 May 28. PMID 24870622
- [Result] Ghia JE, Blennerhassett P, Kumar-Ondiveeran H, Verdu EF, Collins SM. The vagus nerve: a tonic inhibitory influence associated with inflammatory bowel disease in a murine model. Gastroenterology. 2006 Oct;131(4):1122-30. doi: 10.1053/j.gastro.2006.08.016. Epub 2006 Aug 15. PMID 17030182
- [Result] Asconape JJ, Moore DD, Zipes DP, Hartman LM, Duffell WH Jr. Bradycardia and asystole with the use of vagus nerve stimulation for the treatment of epilepsy: a rare complication of intraoperative device testing. Epilepsia. 1999 Oct;40(10):1452-4. doi: 10.1111/j.1528-1157.1999.tb02019.x. PMID 10528943
- [Result] Fahy BG. Intraoperative and perioperative complications with a vagus nerve stimulation device. J Clin Anesth. 2010 May;22(3):213-22. doi: 10.1016/j.jclinane.2009.10.002. PMID 20400010
- [Result] Lacy BE, Patel NK. Rome Criteria and a Diagnostic Approach to Irritable Bowel Syndrome. J Clin Med. 2017 Oct 26;6(11):99. doi: 10.3390/jcm6110099. PMID 29072609
- [Result] Wiklund IK, Fullerton S, Hawkey CJ, Jones RH, Longstreth GF, Mayer EA, Peacock RA, Wilson IK, Naesdal J. An irritable bowel syndrome-specific symptom questionnaire: development and validation. Scand J Gastroenterol. 2003 Sep;38(9):947-54. doi: 10.1080/00365520310004209. PMID 14531531
- [Result] Travers P, Lacy BE, Cangemi DJ. Irritable bowel syndrome - less irritable, or better treatments? Curr Opin Gastroenterol. 2024 Jan 1;40(1):27-33. doi: 10.1097/MOG.0000000000000987. Epub 2023 Oct 19. PMID 38078610

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT06321237/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT06321237/ICF_001.pdf